CLINICAL TRIAL: NCT00532389
Title: A Phase Ib, Multi-center, Open-label, Dose-escalation Study of Oral LBH589 When Administered in Combination With Bortezomib in Adult Patients With Multiple Myeloma
Brief Title: Safety Study of LBH589 When Given in Combination With Bortezomib in Adult Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2207; 2006-006638-16 (EudraCT Number)
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2014-10

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Bortezomib; LBH589; Combination
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Panobinostat

ARMS (1):
- Panobinostat (LBH589) (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589

SUMMARY:
This study comprises of a dose-escalation and dose expansion phase and will determine the maximum tolerated dose of oral Panobinostat on a continuous schedule in adult in combination with bortezomib. Safety, tolerability, PK and PD profile of the combined treatments will be assessed as secondary objectives. Dose expansion phase will explore in a non continuous Panobinostat schedule with bortezomib and dexamethasone, safety and tolerability and PK profile of Panobinostat and Bortezomib with and without Dexamethasone

ELIGIBILITY:
Inclusion criteria:

1. Patients must have a diagnosis of active multiple myeloma according to the International Myeloma Working Group criteria (IMWG., 2003), and be deemed by the investigator as requiring treatment.
2. Patients must have received at least one prior line of therapy and includes patients whose disease has relapsed as well as relapsed-refractory MM . (Durie et. al., 2006). One prior line of therapy may consist of induction followed by autologous stem cell transplantation.
3. Patients must be suitable (according to their local product information and applicable health authority recommendations) for treatment with BTZ. Note: patients previously treated with BTZ are eligible to participate in the trial.
4. Patients enrolled to dose expansion phase must have measurable M component at entry according to the IMWG Criteria (Durie et al, 2006) including at least one of the following:

   * Serum M-protein by sPEP ≥ 1 g/dL (> 10g/l)
   * For patients with IgA M-protein whose sPEP is not providing sufficiently precise quantification due to confounded migration of M-protein with serum beta globulins, a quantification by nephelometry / turbidometry is permitted and must show serum M-protein ≥ 1 g/dL
   * Urine M-protein by uPEP ≥ 200 mg/24 h
   * Serum FLC assay: Involved FLC level ≥ 100 mg/L, provided serum FLC ratio is abnormal. (abnormal if FLC ratio is <0.26 or >1.65 )
5. Adults ≥ 18 years old
6. ECOG Performance Status ≤ 2
7. Life expectancy > 12 weeks
8. Patients must have the following laboratory values:

   * ANC ≥ 1.5 x 109/L
   * Platelets ≥ 100x 109/L
   * Calculated CrCl ≥ 30 mL/min (MDRD Formula)
   * AST and ALT ≤ 2.5 x ULN
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum potassium, magnesium, phosphorous, within normal limits (WNL) for institution
   * Total calcium (corrected for serum albumin) or ionized calcium equal to lower normal limits for institution or greater (≥ LLN) but not higher than CTCAE grade 1
   * Note: Potassium, calcium, magnesium, and/or phosphorous supplements may be given to correct values that are < LLN.
9. Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal
10. All patients (dose-escalation and dose-expansion patients) must be willing to undergo a mandatory bone marrow aspirate sampling at baseline (for cytology) and another later in the study if the patient eventually goes on to experience a CR or PR. For patients who join the study at the dose-expansion phase, they must also give consent to have an extra volume of sample taken for exploratory biomarker testing. Potential dose-expansion phase patients who do not consent for this biomarker sample collection will not be eligible to participate in the trial (Note: One extra bone aspirate sample at C2D1 is optional as per the protocol).
11. Able to sign informed consent and to comply with the protocol
12. Patient is able to swallow capsules

Exclusion criteria:

1. Prior exposure to a HDAC inhibitor compound used in the treatment of MM
2. Patients with Refractory MM (i.e. patients refractory to all prior therapies) who under all prior previous lines of therapy have :

   * either never reached a response better than SD
   * or whose disease progressed from any best response while still under therapy
   * or whose disease progressed within 60 days of last dose of therapy
3. Patients who have had prior allogeneic stem cell transplantation and show evidence of active graft-versus-host disease or of graft-versus-host disease that requires immunosuppressive therapy.
4. Patient has grade 1 peripheral neuropathy with pain or grade ≥ 2 peripheral neuropathy on clinical examination within 14 days before first study treatment
5. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   * Patients with congenital long QT syndrome
   * History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with the Sponsor prior to enrollment)
   * Any history of ventricular fibrillation or torsade de pointes
   * Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
   * Screening ECG with a QTc > 450 msec
   * Right bundle branch block + left anterior hemiblock (bifascicular block)
   * Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
   * Other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
6. Impairment of GI function or GI disease that may significantly alter the absorption of PAN
7. Patient has unresolved diarrhea ≥ CTCAE grade 2
8. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection, acute diffuse pulmonary disease, pericardial disease, uncontrolled thyroid dysfunction ) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
9. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
10. Patients who need valproic acid for any medical condition during the study or within 5 days prior to the first PAN treatment.
11. Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (which ever is longer) and who have not recovered from side effects of those therapies.
12. Patients who have received either immunotherapy within ≤ 8 weeks; chemotherapy within ≤ 4 weeks; or radiation therapy to > 30% of marrow-bearing bone within ≤ 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
13. Patients who have received steroids (e.g. Dex) ≤ 2 weeks prior to starting study treatment or who have not recovered from side effects of such therapy. Concomitant therapy medications that include corticosteroids are allowed if patients receive < 10 mg of prednisone or equivalent as indicated for other medical conditions, or up to 100 mg of hydrocortisone as pre-medication for administration of certain medications or blood products while enrolled in this study.
14. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
15. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP)not willing to use a double method of contraception during the study and for 3 months after treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of oral PAN
16. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and for 3 months after treatment. One of these methods of contraception must be a condom
17. Patients with a prior malignancy with in the last 3 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
18. Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
19. Patients who have shown intolerance to BTZ or to Dex or components of these drugs or has any contraindication to one or the other drug, following locally applicable prescribing information

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To determine the MTD of panobinostat with bortezomib | throughout the study

SECONDARY OUTCOMES:
The safety and tolerability of the study continuous Panobinostat treatment in dose escalation phase and non continuous schedule of panobinostat in dose expansion phase | throughtout the study
To characterize the PK profile of bortezomib; the PK profile of panobinostat with and without bortezomib; the PK profile of bortezomib and panobinostat with and without dexamethasone | cycle 1 & cycle 2
To assess the preliminary efficacy of the study treatment | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (4):
  - Innovative Medical Research of South Florida Dept.ofInnovativeMedResearch, Miami Shores, Florida
  - Dana Farber Cancer Institute Clinical Research Coordinator, Boston, Massachusetts
  - Hackensack University Medical Center Multiple Myeloma Division, Hackensack, New Jersey
  - Swedish Medical Center Dept.ofSwedishMedicalCtr., Seattle, Washington
- Novartis Investigative Site, Canberra, Australian Capital Territory, Australia
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Torino, TO
- Spain (2):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia

REFERENCES:
- See also: Results for CLBH589B2207 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12524